CLINICAL TRIAL: NCT07029477
Title: Incentive Spirometry Versus Massage Therapy on the Level of Shoulder Pain and Nausea Among Post Laparoscopic Cholecystectomy Patients
Brief Title: Incentive Spirometry Versus Massage Therapy Among Post Laparoscopic Cholecystectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sara Arafat Ali Mohamed, Dr, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Spirometry Versus Massage
Record Dates: First submitted 2025-05-25; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Laparoscopic Cholecystectomy; Shoulder Pain; Nausea
MeSH Terms: conditions — Shoulder Pain; Nausea | interventions — Massage

STUDY DESIGN:
Intervention Model Description: quasi-experimental research design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentive Spirometry for Postoperative Pain and Nausea (Experimental): Participants in this group received incentive spirometry therapy only.
  Interventions: Device: Incentive Spirometry
- Massage Therapy for Postoperative Pain and Nausea (Experimental): Participants in this group received massage therapy only.
  Interventions: Behavioral: Massage Therapy

INTERVENTIONS:
Device: Incentive Spirometry — Participants received incentive spirometry therapy using a standard device beginning within 2 hours post-laparoscopic cholecystectomy. They were instructed to take 10 deep breaths every 2 hours for 12 hours.
  Arms: Incentive Spirometry for Postoperative Pain and Nausea
Behavioral: Massage Therapy — Participants received manual massage therapy at regular intervals of 4, 8, and 12 hours after laparoscopic cholecystectomy.
  Arms: Massage Therapy for Postoperative Pain and Nausea

SUMMARY:
The aim of this study is to:

Evaluate the effect of incentive spirometry versus massage therapy on the level of shoulder pain, and nausea among post laparoscopic cholecystectomy patients.

DETAILED DESCRIPTION:
Acute cholecystitis is an inflammation of the gallbladder usually caused by gallstones obstructing the gallbladder neck or cystic duct. It is one of the most common surgical emergency presentations globally. Cholecystectomy was well-known as the surgical care for cholecystitis and the preferred treatment for gallstone disease. Earlier, open cholecystectomy was the gold standard for treatment of cholecystitis. However, open cholecystectomy has been associated with a higher risk of surgical site infection (SSI).

Owing to open surgical procedures complications, the laparoscopic technique has now replaced the open technique in many common surgical procedures, including routine cholecystectomy. Laparoscopic cholecystectomy (LC) is clearly defined as a minimally invasive surgical procedure to remove an inflamed gallbladder resulting from symptomatic cholelithiasis, gallstone, gallbladder masses, or polyps.

Laparoscopic cholecystectomy not only benefits the patient by reducing postoperative pain, discomfort, reducing intraabdominal adhesions, improving cosmetic results, shortening hospital stay, and quickening return to usual activities, but it also benefits the surgeon by improving vision and access to the Calot's triangle. In spite of several blessings of laparoscopic surgical treatment, shoulder pain is considered one of early post laparoscopic symptoms. It seems to have a multifactorial mechanism, but the most reported theory is carbon dioxide gas persistence between the right diaphragm and the hepatic dome that stays inside the abdominal cavity for some times. The surgeon injects CO2 gas into the peritoneum to increase the field of vision dur¬ing cholecystectomy via laparoscopy, this gas causes stretching of the peritoneum and diaphragm, as well as excitation of the phrenic nerve and creation of shoulder pain.

In other words, pain occurs in the scapula through stimulating the phrenic nerve, which originates from the third and fifth cervical nerves (C3-C5) and controls movement and provides sensation in the diaphragm. Postoperative pain can lead to increase heart rate, high blood pressure, and consequently, increase cardiac workload, nausea, vomiting, and ileus.

During laparoscopy, the pneu¬moperitoneum can irritate the vagus nerve, leading to post-operative nausea and vomiting (PONV) which cause delayed discharge, dehydration, wound opening, pulmonary aspiration, patient dissatisfaction, and increased treatment costs. Approximately (50-75%)of patients develop PONV. Prevention and treatment of postoperative pain and control of complications such as nausea and vomiting play an important role in early mobility, improve the quality of surgery, and lead to patient satisfaction, early discharge, and reduce costs.

Pharmacological and non-pharmacological applications are widely used to improve the quality of recovery after laparoscopic cholecystectomy. Pain killers as opioids and nonsteroidal anti-inflammatory drugs have side effects such as respiratory depression, nausea, itching, and bleeding which may affect patient's recovery. Various drugs such as dopamine antagonists, and Dimenhydrinate are used for the prevention and treatment of nausea and vomiting, but each has advantages and disadvantages.

Non-pharmacological nursing measures are cost effective, reduce pain, and analgesic drug dosage, improve patient's emotional control, and increase their functional capability. Variant studies show that shoulder pain is less if the initial pressure of CO2 is maintained below normal levels. With the same approach, chest physiotherapy may have an impact on the mechanical movement of the chest wall and diaphragm. Multiple studies shows and report the dynamic movements of diaphragm and chest wall by cine magnetic resonance image, by stretching the alveoli and chest, the diaphragm's movements increase and contract downward. As a result, less CO2 is accumulated inside the abdominal cavity and result in the removal of CO2.

In this respect, it is essential for surgical nurses to provide education on the proper usage of incentive spirometry to patients, as well as explain its significance and the positive impact of regular intervals on the recovery process. However, studies have found that the rates of teaching and applying deep breathing technique to patients via incentive spirometry are not at the desired level.

Therapeutic massage is also one of the non-pharmacological interventions, it's the manipulation of the soft tissue of whole body areas to bring about generalized improvements in health. It is a non-invasive method with an easy application used to increase the quality of surgery.

The effect of massage on pain is explained with the Gate Control Theory of Melzack. According to this theory, when massage is applied, the A-alpha and A-beta thick tactile fibers moving faster than the A-delta and C fine fibers that are involved in the transmission of the pain, prevent the impulses in the small-diameter fibers that carry the pain from reaching upper levels. The mechanoreceptors that are located in the center of the tactile fibers, which are mentioned in this theory, are found in the hands and feet.

Hand massage has been studied as a potential intervention to reduce postoperative nausea after laparoscopic cholecystectomy. Therefore, the purpose of this study is to evaluate the effect of incentive spirometry versus massage therapy on post laparoscopic cholecystectomy patients in terms of their level of shoulder pain, and nausea.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* Patients aged between 20 to 60 years.
* Patients having the ability to communicate.
* Willing to participate in the study.

Exclusion Criteria:

* Patients who had postoperative bleeding.
* Patients who had postoperative hemodynamic disorders (severe elevation or reduction of blood pressure and shock).
* Patients who had postoperative complications requiring mechanical ventilation.
* Patients who had respiratory aspiration.
* Patients who had a history of drug abuse.
* Patients who had previous shoulder pain chronicity
* Uncooperative patients or patients unable to understand how to use the incentive spirometry device properly.
* Patients whose surgery converted from laparoscopic to open surgery

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain Level & Nausea | Within 12 hours post laparoscopic cholecystectomy
  Change in patient-reported shoulder pain and nausea using a Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain or nausea and 10 indicates the worst possible pain or nausea. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Eid Abdel Moneim, Assist Professor, Study Director — Mansoura University; Wafaa Ismail Shereif, Professor, Study Director — Mansoura University
Locations (1):
- Faculty of Nursing. Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
"Due to the strict confidentiality agreements with participants, individual participant data (IPD) will not be shared. Protecting participant privacy and complying with ethical standards are our top priorities."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT07029477/Prot_SAP_000.pdf